CLINICAL TRIAL: NCT05659017
Title: Study to Identify a Genetic Defect in Subjects With Hyperferritinemia.
Brief Title: Candidate Gene for Hyperferritinemia
Acronym: HyFerr
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Sara Pelucchi, Principal Investigator, University of Milano Bicocca
Other Study IDs: HyFerr
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hyperferritinemia
MeSH Terms: conditions — Hyperferritinemia | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — EDTA vacuette
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Genetic analysis — The DNA will then be analyzed with a custom panel designed ad hoc to study the candidate gene by Next Generation Sequencing according to the protocols of the supplier of the kit.

SUMMARY:
Ferritin is a ubiquitous protein capable of storing iron in the cell cytosol. Stored iron is released and made available for cellular needs by the degradation of ferritin itself. Small amounts of ferritin are present in the blood and consist of ferritin L, a glycosylated form of L called ferritin G, and trace amounts of ferritin H. It is secreted mainly by macrophages, hepatocytes, and lymphoid cells, but most aspects of its secretion remain not fully elucidated. Serum ferritin has broad clinical utility primarily as an indicator of iron stores, so low values of serum ferritin are indicative of a deficient state and high values of iron overload. However, the causes of increased serum ferritin are numerous, in many cases serum ferritin is increased disproportionately to iron stores such as in acute and chronic liver disease, infectious and inflammatory states, metabolic disorders, and high alcohol intake that are frequently observed in the clinical setting. Therefore, the diagnosis of hyperferritinemia requires a careful strategy including personal and family history, biochemical, instrumental, and targeted genetic testing. In fact, there are rare forms of genetically determined hyperferritinemia not associated with iron overload, such as hereditary cataract hyperferritinemia syndrome (HHCS) due to mutations in the Iron responsive Element (IRE) located in the 5' untranslated region of the FTL gene. More recently, a second dominant form of genetic hyperferritinemia without iron overload or cataract (benign hyperferritinemia) has been identified.

Preliminary results obtained so far have made it possible, through WES analysis, to identify the involvement of the STAB1 gene, which was found to be mutated in the studied subjects in whom reduced serum ferritin glycosylation and reduced plasma concentration of the protein itself were observed. It is therefore deemed necessary to proceed with the assay of glycosylated ferritin and the protein encoded by the gene to assess its sensitivity and specificity as a predictive test before performing the genetic analysis of STAB1. To achieve this goal, patients with undefined hyperferritinemia afferent to the SSD Rare Diseases of the IRCCS San Gerardo Foundation in whom to perform glycosylated ferritin and STAB1 protein assay in parallel with STAB1 sequencing will be evaluated. Similar investigations will be performed in a control group consisting of cases of hyperferritinemia due to genetically determined iron overload.

DETAILED DESCRIPTION:
Ferritin is a ubiquitous protein capable of storing iron in the cell cytosol. Cytosolic ferritin consists of two subunits, the light chain (L-ferritin) and the heavy chain (H-ferritin) that assemble in different proportions to form apo-ferritin shells. Ferritin nanoshells consist of 24 subunits of the L- and H-chains that create a cavity in which intracellular iron is collected. The stored iron is released and made available for cellular needs by the degradation of ferritin. Ferritin can bind, oxidize, and store up to 4500 Fe(II) atoms, preventing iron-mediated oxidative stress. This is achieved by regulating ferritin synthesis according to cellular iron content and oxidative stress at both the post-transcriptional (via the Iron Responsive Element (IRE)-regulatory protein (IRP) system) and transcriptional levels. Small amounts of ferritin are present in the blood and consist of ferritin L, a glycosylated form of L called ferritin G, and traces of ferritin H. It is secreted primarily by macrophages, hepatocytes, and lymphoid cells, but most aspects of its secretion remain unknown. Serum ferritin has broad clinical utility primarily as an indicator of intracellular iron stores.

The causes of increased serum ferritin are numerous, including primary and secondary iron overload disorders, but also conditions in which serum ferritin is increased disproportionately to the body's iron stores such as chronic liver disease, inflammatory and metabolic disorders that are frequently observed in the clinical setting. Therefore, the diagnosis of hyperferritinemia requires a systematic strategy including personal and family history, biochemical and instrumental tests. In addition, alterations in the regulation of ferritin synthesis due to mutations in the iron-sensitive element L-ferritin (IRE) cause hereditary hyperferritinemia cataract syndrome (HHCS), an inherited disease characterized by elevated serum ferritin without iron overload and early onset of bilateral cataracts. Recently, a second dominant form of genetic hyperferritinemia without iron overload or cataract has been reported. Amino acid substitutions at positions 26, 27, and 30 in the heterozygous state in the L-ferritin A helix have been found in these patients. The resulting ferritin appears unusually susceptible to glycosylation, leading to serum glycosylated ferritin values consistently >90%. The reason for the development of hyperferritinemia and hyperglycosylation associated with these mutant forms of ferritin has not been established. It is probably related to increased secretion, but may also contribute to delayed clearance. Some cases of hyperferritinemia still remain unexplained, and the currently unknown candidate gene that we think we have identified among candidate genes needs to be validated in a larger population of subjects with the listed characteristics.

The primary objective of the study is to sequence the candidate gene that emerged from previous studies as mutated in patients with the same clinical features.

The secondary objective is to include the candidate gene in the routine genetic diagnosis of subjects with hyperferritinemia without tissue iron overload.

The study will last about 12 months the time needed for the recovery of patients with a genetic diagnosis not yet defined, analysis of medical records and research of the DNA sample stored at the Laboratory of Cytogenetics and Medical Genetics of San Gerardo Hospital and genetic analysis by Next Generation Sequencing. The study, although simple in its idea, requires a very careful organization of access and monitoring of selected patients that require the presence of a study manager dedicated to the project.

The study extension includes:glycosylated ferritin assay in patients with hyperferritinemia referred to the Rare Disease Center of IRCCS Foundation - San Gerardo dei Tintori selected according to the inclusion and exclusion criteria; soluble protein assay encoded by the STAB1 gene in patients in point A and patients in group D.

ELIGIBILITY:
Inclusion Criteria:

Among patients referred to the Center for Rare Diseases of Monza will be enrolled only subjects with:

* ferritin > 1000 g / L in men and > 500 g / L,
* transferrin saturation <45%
* absence of hepatic iron overload, evaluated by liver biopsy or MRI, as indicated in the attached flow chart.

Exclusion Criteria:

Patients with hyperferritinemia attributable to:

* genetically determined causes [mutations in the HFE gene (homozygosity or heterozygosity for p.Cys282Tyr, homozygosity for p.His63Asp or compound heterozygosity for variants of p.Cys282Tyr and p. His63Asp), ferroportin and L-Ferritin gene mutations];
* presence of more than one component of metabolic syndrome (according to NCEP-ATPIII criteria: triglycerides >150 mg/dL, blood glucose >100 mg/dL, HDL <40 mg/dL in men and <50 mg/dL in women, waist circumference >102 cm in men and >88 cm in women; blood pressure ≥130/≥85 mm/Hg);
* alcohol intake >5 g/day chronic hepatitis,
* history of blood transfusion or parenteral iron treatment,
* late skin porphyria,
* hyperthyroidism,
* presence of cataracts or family history of early-onset cataracts
* acute or chronic inflammatory disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hyperferritinemia patients followed at the Rare Diseases Center in San Gerardo Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Candidate gene sequencing | 1 year
  For the purpose 100 patients are sufficient to calculate both the allelic and genotypic frequency of mutations in the candidate gene.

SECONDARY OUTCOMES:
DIAGNOSIS ROUTINE | 1 year
  The secondary objective is to include the candidate gene in the routine genetic diagnosis of individuals with hyperferritinemia without tissue iron overload.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Rare Disease - Disorders of Iron Metabolism, ASST-Monza, San Gerardo Hospital, European Reference Network - EuroBloodNet, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arosio P, Levi S. Cytosolic and mitochondrial ferritins in the regulation of cellular iron homeostasis and oxidative damage. Biochim Biophys Acta. 2010 Aug;1800(8):783-92. doi: 10.1016/j.bbagen.2010.02.005. Epub 2010 Feb 20. PMID 20176086
- [Result] Torti FM, Torti SV. Regulation of ferritin genes and protein. Blood. 2002 May 15;99(10):3505-16. doi: 10.1182/blood.v99.10.3505. No abstract available. PMID 11986201
- [Result] Finazzi D, Arosio P. Biology of ferritin in mammals: an update on iron storage, oxidative damage and neurodegeneration. Arch Toxicol. 2014 Oct;88(10):1787-802. doi: 10.1007/s00204-014-1329-0. Epub 2014 Aug 15. PMID 25119494
- [Result] Wang J, Pantopoulos K. Regulation of cellular iron metabolism. Biochem J. 2011 Mar 15;434(3):365-81. doi: 10.1042/BJ20101825. PMID 21348856
- [Result] Cragg SJ, Wagstaff M, Worwood M. Sialic acid and the microheterogeneity of human serum ferritin. Clin Sci (Lond). 1980 Mar;58(3):259-62. doi: 10.1042/cs0580259. PMID 7363568
- [Result] Santambrogio P, Cozzi A, Levi S, Arosio P. Human serum ferritin G-peptide is recognized by anti-L ferritin subunit antibodies and concanavalin-A. Br J Haematol. 1987 Feb;65(2):235-7. doi: 10.1111/j.1365-2141.1987.tb02271.x. PMID 3828232
- [Result] Cohen LA, Gutierrez L, Weiss A, Leichtmann-Bardoogo Y, Zhang DL, Crooks DR, Sougrat R, Morgenstern A, Galy B, Hentze MW, Lazaro FJ, Rouault TA, Meyron-Holtz EG. Serum ferritin is derived primarily from macrophages through a nonclassical secretory pathway. Blood. 2010 Sep 2;116(9):1574-84. doi: 10.1182/blood-2009-11-253815. Epub 2010 May 14. PMID 20472835
- [Result] Mack U, Cooksley WG, Ferris RA, Powell LW, Halliday JW. Regulation of plasma ferritin by the isolated perfused rat liver. Br J Haematol. 1981 Mar;47(3):403-12. doi: 10.1111/j.1365-2141.1981.tb02808.x. PMID 7459278
- [Result] Tran TN, Eubanks SK, Schaffer KJ, Zhou CY, Linder MC. Secretion of ferritin by rat hepatoma cells and its regulation by inflammatory cytokines and iron. Blood. 1997 Dec 15;90(12):4979-86. PMID 9389717
- [Result] Dorner MH, Silverstone A, Nishiya K, de Sostoa A, Munn G, de Sousa M. Ferritin synthesis by human T lymphocytes. Science. 1980 Aug 29;209(4460):1019-21. doi: 10.1126/science.6967622.
- [Result] Byg KE, Milman N, Hansen S, Agger AO. Serum Ferritin is a Reliable, Non-invasive Test for Iron Status in Pregnancy: Comparison of Ferritin with Other Iron Status Markers in a Longitudinal Study on Healthy Pregnant Women; Erythropoiesis. Hematology. 2000;5(4):319-325. doi: 10.1080/10245332.2000.11746526. PMID 11399631
- [Result] Harrison PM, Arosio P. The ferritins: molecular properties, iron storage function and cellular regulation. Biochim Biophys Acta. 1996 Jul 31;1275(3):161-203. doi: 10.1016/0005-2728(96)00022-9. PMID 8695634
- [Result] Jacobs A, Worwood M. Ferritin in serum. Clinical and biochemical implications. N Engl J Med. 1975 May 1;292(18):951-6. doi: 10.1056/NEJM197505012921805. No abstract available. PMID 1090831
- [Result] Chen TT, Li L, Chung DH, Allen CD, Torti SV, Torti FM, Cyster JG, Chen CY, Brodsky FM, Niemi EC, Nakamura MC, Seaman WE, Daws MR. TIM-2 is expressed on B cells and in liver and kidney and is a receptor for H-ferritin endocytosis. J Exp Med. 2005 Oct 3;202(7):955-65. doi: 10.1084/jem.20042433. PMID 16203866
- [Result] Li JY, Paragas N, Ned RM, Qiu A, Viltard M, Leete T, Drexler IR, Chen X, Sanna-Cherchi S, Mohammed F, Williams D, Lin CS, Schmidt-Ott KM, Andrews NC, Barasch J. Scara5 is a ferritin receptor mediating non-transferrin iron delivery. Dev Cell. 2009 Jan;16(1):35-46. doi: 10.1016/j.devcel.2008.12.002. PMID 19154717
- [Result] Ravasi G, Pelucchi S, Mariani R, Casati M, Greni F, Arosio C, Pelloni I, Majore S, Santambrogio P, Levi S, Piperno A. Unexplained isolated hyperferritinemia without iron overload. Am J Hematol. 2017 Apr;92(4):338-343. doi: 10.1002/ajh.24641. Epub 2017 Feb 7. PMID 28052375
- [Result] Aguilar-Martinez P, Schved JF, Brissot P. The evaluation of hyperferritinemia: an updated strategy based on advances in detecting genetic abnormalities. Am J Gastroenterol. 2005 May;100(5):1185-94. doi: 10.1111/j.1572-0241.2005.40998.x. PMID 15842597
- [Result] Camaschella C, Poggiali E. Towards explaining "unexplained hyperferritinemia". Haematologica. 2009 Mar;94(3):307-9. doi: 10.3324/haematol.2008.005405. PMID 19252171
- [Result] Kannengiesser C, Jouanolle AM, Hetet G, Mosser A, Muzeau F, Henry D, Bardou-Jacquet E, Mornet M, Brissot P, Deugnier Y, Grandchamp B, Beaumont C. A new missense mutation in the L ferritin coding sequence associated with elevated levels of glycosylated ferritin in serum and absence of iron overload. Haematologica. 2009 Mar;94(3):335-9. doi: 10.3324/haematol.2008.000125. Epub 2009 Jan 27. PMID 19176363
- [Result] Thurlow V, Vadher B, Bomford A, DeLord C, Kannengiesser C, Beaumont C, Grandchamp B. Two novel mutations in the L ferritin coding sequence associated with benign hyperferritinaemia unmasked by glycosylated ferritin assay. Ann Clin Biochem. 2012 May;49(Pt 3):302-5. doi: 10.1258/acb.2011.011229. Epub 2012 Apr 25. PMID 22535864
- [Result] Piperno A. Molecular diagnosis of hemochromatosis. Expert Opin Med Diagn. 2013 Mar;7(2):161-77. doi: 10.1517/17530059.2013.763794. Epub 2013 Jan 23. PMID 23530886
- [Result] Riva A, Trombini P, Mariani R, Salvioni A, Coletti S, Bonfadini S, Paolini V, Pozzi M, Facchetti R, Bovo G, Piperno A. Revaluation of clinical and histological criteria for diagnosis of dysmetabolic iron overload syndrome. World J Gastroenterol. 2008 Aug 14;14(30):4745-52. doi: 10.3748/wjg.14.4745. PMID 18720534
- [Result] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966